CLINICAL TRIAL: NCT01746134
Title: A Prospective, Non-Interventional Registry of Diverse Patients With Schizophrenia Across the Disease Spectrum in Usual Care Settings: Course of Disease, Treatments, and Burden of Illness
Brief Title: The Management of Schizophrenia in Clinical Practice (MOSAIC)
Status: Completed | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28264
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This study is a disease-based registry designed to follow patients with a DSM-IV-TR (Diagnostic and Statistic Manual of Mental Disorders, Text Revision) diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder treated in usual care settings for up to 5 years. The registry seeks to describe the course of disease in schizophrenia, including cognitive function and negative symptoms, its treatment, and its burden of disease for participants, caregivers, clinicians, and society as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* DSM-IV-TR diagnosis of schizophrenia, schizoaffective disorder, or schizophreniform disorder
* Participants presenting with the normal course of care in usual treatment settings
* Able to read and speak English
* Able and willing to provide informed consent
* Able and willing to comply with the study protocol

Exclusion Criteria:

* Participants enrolled as subjects in clinical trials at registry enrollment
* Participants anticipating they will be unable to participate in regularly scheduled assessments as per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with schizophrenia, schizoaffective disorder, or schizophreniform across the disease spectrum treated in usual care settings
Sampling Method: Probability Sample
Enrollment: 557 (Actual)
Dates: Start 2012-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Symptoms of Schizophrenia (PANSS) | up to 5 years
Clinical Global Impression Schizophrenia Scale (CGI-SCH) | up to 5 years
Cognitive function (Fluency, Digit Symbol-Coding, Trail Making Test) | up to 5 years

SECONDARY OUTCOMES:
Negative Symptom Assessment Scale (NSA4) | up to 5 years
Pharmacologic/behavioural treatments used in usual care settings: intervention | up to 5 years
Pharmacologic/behavioural treatments used in usual care settings: dose | up to 5 years
Pharmacologic/behavioural treatments used in usual care settings: duration | up to 5 years
Personal and Social Performance (PSP) | up to 5 years
Schizophrenia Quality of Life Scale (SQLS) | up to 5 years
Schizophrenia Caregiver Questionnaire | up to 5 years
Maslach Burnout Inventory (MBI) | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (30):
- United States (30):
  - Granada Hills, California
  - Los Angeles, California
  - Santa Monica, California
  - Cedar Rapids, Connecticut
  - New Haven, Connecticut
  - Chicago, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lake City, Florida
  - Miami, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Belmont, Massachusetts
  - Minneapolis, Minnesota
  - Saint Paul, Minnesota
  - New York, New York
  - Orangeburg, New York
  - Carrboro, North Carolina
  - Cary, North Carolina
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Hillsborough, North Carolina
  - Pinehurst, North Carolina
  - Cincinnati, Ohio
  - Lytle, Texas
  - Round Rock, Texas
  - San Antonio, Texas
  - Taylor, Texas
  - Salt Lake City, Utah
  - Tacoma, Washington